CLINICAL TRIAL: NCT00516191
Title: A Phase I/II Study of Liposomal Doxorubicin (Doxil)/Melphalan/Bortezomib (Velcade) in Relapsed/Refractory Multiple Myeloma
Acronym: DMV
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Thomas Martin, MD, Assistant Clinical Professor Medicine, University of California San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-2408
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Velcade; Doxil; Melphalan
MeSH Terms: conditions — Multiple Myeloma | interventions — liposomal doxorubicin; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Liposomal Doxorubicin/Melphalan/Bortezomib — Day 1 Bortezomib 0.7 mg/m(2)IV + Doxil 10-20 mg/m(2)IV+Melphalan 5-10mg/m(2)IV Day 4 Bortezomib 0.7 mg/m(2)IV Day 8 Bortezomib 0.7 mg/m(2)IV Day 11 Bortezomib 0.7 mg/m(2)IV
  The treatment cycles will be repeated every 28 days. Dose Level 1: Doxil 10mg/m(2), Melphalan 5 mg/m(2), Bortezomib 0.7mg/m(2) Dose Level 2: Doxil 10mg/m(2), Melphalan 10 mg/m(2), Bortezomib 0.7mg/m(2) Dose Level 3: Doxil 20mg/m(2), Melphalan 10 mg/m(2), Bortezomib 0.7mg/m(2) Dose Level 4: Doxil 20mg/m(2), Melphalan 10 mg/m(2), Bortezomib 1.0mg/m(2)
  Other Names: Liposomal Doxorubicin=Doxil; Melphalan=Alkeran; Bortezomib=Velcade

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of four dose levels of liposomal doxorubicin, melphalan, and bortezomib in patients with relapsed/refractory MM and to identify a maximum tolerated dose (MTD) of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with multiple myeloma; Durie-Salmon Stage I, II, or III based on standard criteria
* Progressive disease, defined as 25% increase in serum M-protein or Bence Jones protein (an absolute increase of 0.5 gram/dL serum M-protein or at least 200 mg/24 hours of urine light chain excretion). For non-secretory multiple myeloma, progressive disease is defined as bone marrow biopsy with >25% increase in plasma cells or an absolute increase of at least 10% over prior known level. Alternatively, development of new or worsening of existing lytic bone lesions or soft tissue plasmacytomas, or hypercalcemia or relapse from CR.
* 18 year or older and willing and able to comply with the protocol requirements.
* Patient has signed informed consent.
* Unless a female patient is post-menopausal or surgically sterilized, must be willing to use an acceptable method of birth control (hormonal contraceptive, intrauterine device, diaphragm, with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient must agree to use an acceptable method for contraception for the duration of the study.
* ECOG performance Status of < or equal to 2.
* Life expectancy is at least 3 months.
* Initial Required Laboratory Values within 14 days of baseline i.e. Cycle 1, Day 1 (note that renal insufficiency, including dialysis dependence is permissable):

  * ANC>1,000uL without the use of colony stimulating factors
  * Platelets >50,000/L without transfusion support 7 days before the test
  * Bilirubin < or equal to 2.0 mg/dL
  * AST < or equal to 4 x upper limit of normal
* Prior therapy: Patient must have had at least 2 prior therapeutic regimens as defined below for treatment of multiple myeloma

  * Biologic therapy:
* Prior nonmyeloablative transplantation allowed provided patient does not have significant graft-versus-host disease and is off aggressive immunosuppressive therapy for at least 30 days. Low dose immunosuppression is allowed (i.e. Prednisone at dose < or equal to 10 mg daily, low dose tacrolimus (subtherapeutic levels) or other agents with equivalent low-dose immunosuppression).

  * Chemotherapy:
* Mobilization with chemotherapy followed by either single or tandem autologous transplantation is counted as 1 prior regimen.
* Mobilization with chemotherapy followed by autologous and subsequent nonmyeloablative allogenic transplantation is counted as 1 prior regimen.
* Any combination of drugs given concurrently is counted as a single regimen.

Exclusion Criteria:

* Pregnant or breast-feeding
* History of allergic reaction to compounds containing boron or mannitol.
* Active uncontrolled viral (including HIV), bacterial, or fungal infection.
* Grade III or IV toxicity due to previous anti-neoplastic therapy (except alopecia).
* Grade > or equal to 2 motor or sensory neuropathy as defined by the NCI Common Toxicity Criteria (NCI CTC):
* Grade 2: Either mild objective weakness or objective sensory loss/parasthesia (including tingling) that interferes with function, but not interfering with ADLs.
* Grade 3: Objective weakness or sensory loss/parasthesia interfering with ADLs.
* Grade 4: Paralysis or permanent sensory loss that interferes with function.
* Myocardial infarction within 6 months of enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled arrhythmias, or electrocardiographic evidence of acute ischemia.
* For any patients whose lifetime cumulative doxorubicin dose exceeds 400 mg/m(2), patients with LVEF < or equal to 35% by MUGA are excluded. In other patients, MUGA is not required but if performed, LVEF must be > or equal to 35%.
* Concurrent administration of liposomal doxorubicin, melphalan, and bortezomib (single or two drug combinations of these are permissable).
* Less than 3 weeks since most recent chemotherapy or concurrent chemotherapy.
* Use of corticosteroids (>10 mg prednisone/day or equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
--To evaluate the safety and tolerability of four dose levels of liposomal doxorubicin, melphalan, and bortezomib in patients with relapsed/refractory MM and to identify a maximum tolerated dose of this combination. | 6 years

SECONDARY OUTCOMES:
--To determine the efficacy of DMV therapy --Tabulate all the toxicities of DMV at the MTD by NCI criteria | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Cancer Center Home Page — http://cancer.ucsf.edu